CLINICAL TRIAL: NCT01154530
Title: Chlorhexidine Mouthwash and Bacterial Contamination During Endoscopy. Implementation of Chlorhexidine Mouthwash Before Transgastric NOTES
Brief Title: Chlorhexidine Mouthwash and Bacterial Contamination During Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Anders Meller Donatsky, MD, resident, Phd-student, Herlev Hospital, Department of surgical gastroenterology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NOTES01
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2010-12

CONDITIONS: Gastroscopy
Keywords: Gastroscopy; Bacteria; Chlorhexidine; General surgery
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine mouthwash (Active Comparator): Participants randomized to chlorhexidine mouthwash prior to gastroscopy
  Interventions: Other: Chlorhexidine
- No mouthwash (No Intervention): Mouthwash is not performed prior to gastroscopy as is the standard today.

INTERVENTIONS:
Other: Chlorhexidine — Mouthwash with a 0,2 % chlorhexidine solution for 30 seconds
  Arms: Chlorhexidine mouthwash

SUMMARY:
Background:

Natural Orifice Transluminal Endoscopic Surgery (NOTES) is a surgical technique that has been rapidly evolving over the last five years. The technique probably has a great potential in surgical gastroenterology, urology and gynaecology.

The technique is based on the idea of minimally invasive surgery. The human organism is affected by a stress response when exposed to surgery. This stress response can be minimized by reducing the size of the openings whereby the surgeon gains access to the organs. This affects how quickly a patient recovers after surgery and can be discharged and resumes daily life and work. The same principal have been responsible for the surgical evolution in the last 15-20 years where many procedures have gone from traditional open operations with large incisions in the abdominal wall to laparoscopic surgery with cameras through small holes in the abdominal wall.

The latest addition to minimal invasive surgery is NOTES. Here the surgeon gains access to the abdominal organs with flexible endoscopes through the body's natural openings i.e. the mouth and stomach. With this technique the surgeon avoids cutting through skin and muscle of the abdominal wall, thus minimizing the surgical stress response. This minimizes postoperative pain, the incidence of incisional hernias, eliminates wound infection, and properly prevents scar tissue formation inside the abdominal cavity which way lead to ileus. The end result is a quicker discharge and a better cosmetic result.

It has been shown in numerous animal studies that NOTES is feasible and in recent years a rapidly increasing number of published patient series.

However, there is a risk of infection associated with accessing the abdominal cavity through a natural body opening, which initially is unclean and can not be disinfected in the same way as the skin of the abdominal wall.

Numerous microbiological pig studies have shown that there is transfer of bacteria from the body opening (i.e. mouth) to the abdominal cavity when performing NOTES, but this contamination have no correlation to infection after surgery, neither in terms of healing or survival.

It is unclear from the literature whether patients should be offered proton pump inhibitor (PPI) therapy to reduce the acidity of the stomach before NOTES interventions. The rationale has been that such a treatment can make the gastric juices less acidic and thereby reduce the incidence of chemical peritonitis, which can occur when acidic juices flows from the stomach and into the abdominal cavity. It is known however that the acidic environment of the stomach provides a natural barrier for bacteria. Making the gastric juices less acidic could potentially increase the risk of bacterial peritonitis.

It is known that the bacterial content of the stomach is low due the acidic environment but bacteria passed down from the mouth and throat with the endoscope could potentially result in bacterial peritonitis.

That bacteria from the throat can lead to infections due to instrumentation is known from intensive care units. Ventilated patients may risk getting pneumonia with bacteria from the throat. Several studies have shown that using mouthwash with a chlorhexidine solution can reduce the risk of ventilator associated pneumonia.

Hypothesis:

Mouthwash with 2 cl 0,2% chlorhexidine solution before a gastroscopy reduces the bacterial content in cultures taken from the stomach and the endoscope after a gastroscopy.

Simultaneous PPI treatment gives higher bacterial counts in the cultures.

DETAILED DESCRIPTION:
Background:

Natural Orifice Transluminal Endoscopic Surgery (NOTES) is a surgical technique that has been rapidly evolving over the last five years. The technique probably has a great potential in surgical gastroenterology, urology and gynaecology.

The technique is based on the idea of minimally invasive surgery. The human organism is affected by a stress response when exposed to surgery. This stress response can be minimized by reducing the size of the openings whereby the surgeon gains access to the organs. This affects how quickly a patient recovers after surgery and can be discharged and resumes daily life and work. The same principal have been responsible for the surgical evolution in the last 15-20 years where many procedures have gone from traditional open operations with large incisions in the abdominal wall to laparoscopic surgery with cameras through small holes in the abdominal wall.

The latest addition to minimal invasive surgery is NOTES. Here the surgeon gains access to the abdominal organs with flexible endoscopes through the body's natural openings i.e. the mouth and stomach. With this technique the surgeon avoids cutting through skin and muscle of the abdominal wall, thus minimizing the surgical stress response. This minimizes postoperative pain, the incidence of incisional hernias, eliminates wound infection, and properly prevents scar tissue formation inside the abdominal cavity which way lead to ileus. The end result is a quicker discharge and a better cosmetic result.

It has been shown in numerous animal studies that NOTES is feasible and in recent years a rapidly increasing number of published patient series.

However, there is a risk of infection associated with accessing the abdominal cavity through a natural body opening, which initially is unclean and can not be disinfected in the same way as the skin of the abdominal wall.

Numerous microbiological pig studies have shown that there is transfer of bacteria from the body opening (i.e. mouth) to the abdominal cavity when performing NOTES, but this contamination have no correlation to infection after surgery, neither in terms of healing or survival.

It is unclear from the literature whether patients should be offered proton pump inhibitor (PPI) therapy to reduce the acidity of the stomach before NOTES interventions. The rationale has been that such a treatment can make the gastric juices less acidic and thereby reduce the incidence of chemical peritonitis, which can occur when acidic juices flows from the stomach and into the abdominal cavity. It is known however that the acidic environment of the stomach provides a natural barrier for bacteria. Making the gastric juices less acidic could potentially increase the risk of bacterial peritonitis.

It is known that the bacterial content of the stomach is low due the acidic environment but bacteria passed down from the mouth and throat with the endoscope could potentially result in bacterial peritonitis.

That bacteria from the throat can lead to infections due to instrumentation is known from intensive care units. Ventilated patients may risk getting pneumonia with bacteria from the throat. Several studies have shown that using mouthwash with a chlorhexidine solution can reduce the risk of ventilator associated pneumonia.

Hypothesis:

Mouthwash with 2 cl 0,2% chlorhexidine solution before a gastroscopy reduces the bacterial content in cultures taken from the stomach and the endoscope after a gastroscopy.

Simultaneous PPI treatment gives higher bacterial counts in the cultures.

Trial Participants:

Trial Participants will be recruited among patients referred to gastroscopy in an outpatient setting, at Herlev, Gentofte and Bispebjerg Hospital.

Participants must be over 18 years old regardless of gender. The participants are included after oral and written information about the trial and with written consent. The request for participation and written information about the trial is send to the patient by conventional mail. The oral information is given on the day of the gastroscopy. Inclusion in the trial has no consequences for the purpose of the gastroscopy, or on any further diagnostic procedures or treatments. Trial Participants may at any time withdraw from the trial without consequences.

Method:

Included participants are randomized by drawing a random envelope with a continuous registration number containing information on whether the patient is allocated to the intervention or control group.

Enclosed in the envelope is a registration form where the following is recorded: sex, age, weight, height, indication for gastroscopy, number of instrumentations during gastroscopy, the use of rinse and suction, and PPI treatment.

Participants in the intervention group perform a mouthwash with 2 cl 0,2% chlorhexidine for 30 seconds immediately before the gastroscopy.

Participants in the control group perform no mouthwash before the gastroscopy.

The gastroscopy is performed in accordance with the indication.

A total of 2 culture samples will be taken from each participant. The culture samples are sent to the department of clinical microbiology, Herlev Hospital for cultivation, bacterial count and typing.

The first culture sample is taken by instilling 50ml sterile saline through the instrumentation channel with the gastroscope located in the fundus of the stomach . Approximately 10ml is aspirated through the same channel in the antrum of the stomach.

The second culture sample is taken from the gastroscope after the procedure by rinsing the instrumentation channel with sterile saline. A sample of approximately 10 ml is collected at the distal end of the gastroscope.

Samples are marked with the respective continuous registration numbers according to the randomization.

Side effects, discomfort and risks:

There are no side effects associated with the use chlorhexidine mouthwash.

There is some discomfort associated with the gastroscopy. This is not a result of participation in the trial.

Many patients feel slight discomfort when the gastroscope passes through the throat. The passage can stimulate the vomiting reflex. For this reason a gastroscopy is always performed with the patient in a left lateral position to ensure free airways. There may be mild soreness and irritation in the throat during and in the first few days after the gastroscopy.

The only discomfort that is directly linked to participation in the trial is the taste of chlorhexidine mouthwash for half of the participants.

There are no risks associated with participation in the trial, although there are some risks associated with the gastroscopy itself. These are bleeding from the stomach wall and perforation of the stomach or duodenum. These complications are very rare.

Ethics:

Since the participants are recruited after referral to gastroscopy from a general practitioner the indication for the gastroscopy has already been assessed and outweighs the above mentioned rare risks.

The only discomfort that is directly related to the trail is a brief sensation of bad taste in the mouth for half of the participants.

The results gained from the trial greatly overshadow the mild discomfort associated with the taste of chlorhexidine mouthwash.

Economy:

The above mentioned trial is a part of a PhD project which tries to bridge the gap between animal studies and the implementation of NOTES in daily clinical practice.

Salaries are funded through grants from the University of Copenhagen, Herlev Hospital Research Council and the Capitol Region of Denmark Research Foundation for Health Research. Operating costs are founded through grants from private foundations. There is no commercial interest in or support for the project.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 18 years referred to gastroscopy in an outpatient setting.
* Danish speaking.
* Written informed consent after verbal and written information.

Exclusion Criteria:

* Feeding tube, or the use of a gastric or duodenal tube in the week prior to inclusion.
* Gastroscopy in the week prior to inclusion.
* Removable prosthetic teeth.
* Use of antiseptic mouthwash in the week prior to inclusion.
* Gastroenteroanastomosis.
* Gastrocystotomy.
* Stents in oesophagus / stomach / duodenum / pancreatic or hepatic ducts.
* Known cancer in esophagus / stomach / duodenum / pancreas.
* Percutaneous Endoscopic Gastrostomy / Percutaneous Ultrasonic Gastrostomy
* Known infection or in antibiotic treatment.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Quantification of culture samples | 1 week
  Bacterial count in the culture samples. Quantified with colony forming units (CFU).

SECONDARY OUTCOMES:
The influence of PPI treatment on bacterial count | 1 week
  To study whether ongoing PPI treatment gives higher bacterial counts in the culture samples
Bacteria species | 1 week
  Classification of bacteria species in the culture samples

CONTACTS AND LOCATIONS:
Overall Officials: Anders Meller Donatsky, MD, Principal Investigator — Herlev Hospital, Department of surgical gastroenterology; Jacob Rosenberg, MD DSc Prof, Study Director — Herlev Hospital, Department of surgical gastroenterology; Søren Meisner, MD, Study Director — Bispebjerg Hospital, Department of surgical gastroenterology; Lars Nannestad Jørgensen, MD DSc prof, Study Director — Bispebjerg Hospital, Department of surgical gastroenterology; Peter Vilmann, MD DSc Prof, Study Director — Gentofte Hospital, Department of surgical gastroenterology
Locations (1):
- Herlev Hospital, Department of surgical gastroenterology, Herlev, Denmark